CLINICAL TRIAL: NCT04209790
Title: Phase II Study of Neoadjuvant Chemoradiation for Resectable Glioblastoma (NeoGlio)
Brief Title: Neoadjuvant Chemoradiation for Resectable Glioblastoma
Acronym: NeoGlio
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Suspended to identify a permanent PI at site level. Decision to Terminate was made on 7/29/25 because no other PI able to take on project.
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0623
Record Dates: First submitted 2019-12-17; First posted 2019-12-24 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma; Surgery; High Grade Glioma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Neoadjuvant Therapy; Drug Therapy; Temozolomide; Benzolamide; Standard of Care

STUDY DESIGN:
Intervention Model Description: After standard treatment of Glioblastoma multiforme (GBM) with resection and adjuvant therapy, local failure the dominant pattern of failure. Neo adjuvant therapy consistently provides the potential for improved local control and removal of residual stem cell niches. The hypothesis is that earlier institution of neo adjuvant chemo radiation therapy in GBM would improve local control and potentially overall survival.
  Involved field radiation is often employed to treat unresectable or sub totally resected GBM. Radiating native GBM is not uncommon as many tumors are not safely resectable due to its location in eloquent brain. Planned neoadjuvant chemo radiation prior to immediate surgical resection in glioblastoma is a novel approach in resectable tumors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemoradiation and surgical resection (Other): The experimental part of the study would be this selection of resectable patients and sequencing neoadjuvant chemoradiation prior to surgery.
  Interventions: Radiation: Neoadjuvant chemoradiation; Drug: Drug Therapy with Temozolomide (benzolamide) (Standard of Care); Procedure: Surgery post Radiation and Temozolomide (benzolamide)

INTERVENTIONS:
Radiation: Neoadjuvant chemoradiation — Intensity modulation radiation therapy (IMRT) with a simultaneous integrated boost with Fixed-gantry IMRT, helical tomotherapy, or Vesicular Modulated Arc Therapy (VMAT) can be used. All photon treatments shall be delivered with megavoltage machines of a minimum energy of 6 Megavolt (MV) photons. Selection of the appropriate photon energy(ies) should be based on optimizing the radiation dose distribution within the target volume and minimizing dose to non-target normal tissue.
  Other Names: Standard adjuvant therapy
Drug: Drug Therapy with Temozolomide (benzolamide) (Standard of Care) — During Concomitant Radiation Therapy on the same day as the first fraction of radiotherapy. Temozolomide will be administered continuously from day 1 of radiotherapy to the last day of radiation at a daily oral dose of 75 mg/m2 for a maximum of 49 days. The drug will be administered orally daily during radiotherapy, as best tolerated by the patient. During weekends without radiotherapy (Saturday and Sunday), the drug will be taken in the morning. The dose will be determined using actual body surface area (BSA) as calculated in square meters at the beginning of the concomitant treatment. The BSA will be calculated from the height obtained at the pretreatment visit. Capsules of temozolomide are available in 5, 20, 100, 140, 180, and 250 mg. The daily dose will be rounded to the nearest 5 mg.
  Other Names: Neoadjuvant therapy
Procedure: Surgery post Radiation and Temozolomide (benzolamide) — Surgical resection of GBM will be done after radiation and Temozolomide treatment.

SUMMARY:
Preoperative therapy has not been well studied in resectable glioblastoma. This study attempts to prospectively assess the feasibility and efficacy of preoperative chemo radiation in improving local control, as this is the predominant mode of failure in these patients leading to poor outcomes.

This Phase II study design would be used to proceed with the study treatment after meeting pre-specified events in the initial phase, with goal being to determine whether the new treatment paradigm is sufficiently promising to warrant a major controlled clinical evaluation against the standard therapy.

DETAILED DESCRIPTION:
Neo adjuvant, preoperative chemo radiation has consistently shown improvements in local disease control or organ preservation in many cancers including head and neck, esophageal, rectal, bladder cancers and sarcomas, leading to improvements in overall survival and limb or organ preservation.

This interventional study will be done in two phases using the Simon two-stage Phase II study design. The median progression-free survival of these patients with current standard of care therapy is in the range of 6-8 months (6.9 months in the standard of care). With the proposed trial of surgical resection of the tumor after chemotherapy and radiation the median progression free survival is anticipated to be approximately 11-12 months from subset analysis of available literature and based on prior data on other disease sites. In other words, the 7-month local progression rates is anticipated to decrease from 50% to 25%, or progression free survival improve from 50-75%

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed GBM with histopathological confirmation.
2. Surgically suitable for subtotal or gross total resection as determined by central review.
3. Karnofsky Performance Status (KPS)>70
4. No contraindication for chemoradiation.
5. Complete blood count (CBC)/differential obtained within 28 days prior to registration, with adequate bone marrow function defined as follows:

   1. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
   2. Platelets ≥ 100,000 cells/mm3;
   3. Hemoglobin ≥ 8.0 g/dl (Note: the use of transfusion or other intervention to achieve Hgb ≥8.0 g/dl is acceptable)
6. Adequate hepatic function within 28 days prior to registration, as defined below:

   1. Alanine Aminotransferase (ALT) and Aspartate transaminase (AST) ≤ 3 x ULN
   2. Bilirubin ≤ 1.5 upper limit of normal (ULN)
7. Negative serum pregnancy test obtained for females of child-bearing potential within 28 days prior to step 2 registration.
8. Ability to get multiplanar contrast enhanced Magnetic Resonance Imaging (MRI)

Exclusion Criteria:

1. Recurrent, unresectable or multifocal malignant gliomas.
2. Any site of distant disease (for example, drop metastases from the GBM tumor site)
3. Prior radiation or chemotherapy or radiosensitizers for cancers of the brain and head and neck region; note that prior chemotherapy for a different cancer is allowable (except temozolomide).
4. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
5. Patents treated on any other therapeutic clinical protocols within 30 days prior to registration.
6. Inability to undergo MRI (e.g., due to safety reasons, such as presence of a pacemaker, or severe claustrophobia).
7. Severe, active co-morbidity, defined as follows:

   1. Transmural myocardial infarction within the last 6 months prior to registration
   2. History of recent myocardial infarction 1month prior
   3. New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 3 months prior to registration.
   4. Serious or non-healing wound, ulcer or bone fracture or history of abdominal fistula, intra-abdominal abscess requiring major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to registration, with the exception of the craniotomy for surgical resection
   5. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   6. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol.
   7. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   8. Acquired immune deficiency syndrome (AIDS) based upon current Center for Disease Control (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is because the treatments involved in this protocol may be significantly immunosuppressive with potentially fatal outcomes in patients already immunosuppressed.
   9. Any other severe immuno-compromised condition.
   10. Active connective tissue disorders, such as lupus or scleroderma that in the opinion of the treating physician may put the patient at high risk for radiation toxicity.
   11. End-stage renal disease (i.e. on dialysis or dialysis has been recommended).
   12. Any other major medical illnesses or psychiatric treatments that in the investigator's opinion will prevent administration or completion of protocol therapy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Lacroix, M.D., Principal Investigator — Geisinger Clinic
Locations (2):
- United States (2):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milano MT, Okunieff P, Donatello RS, Mohile NA, Sul J, Walter KA, Korones DN. Patterns and timing of recurrence after temozolomide-based chemoradiation for glioblastoma. Int J Radiat Oncol Biol Phys. 2010 Nov 15;78(4):1147-55. doi: 10.1016/j.ijrobp.2009.09.018. Epub 2010 Mar 6. PMID 20207495
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Yarbro JW. Future potential of adjuvant and neoadjuvant therapy. Semin Oncol. 1991 Dec;18(6):613-9. No abstract available. PMID 1775978
- [Background] Filatova A, Acker T, Garvalov BK. The cancer stem cell niche(s): the crosstalk between glioma stem cells and their microenvironment. Biochim Biophys Acta. 2013 Feb;1830(2):2496-508. doi: 10.1016/j.bbagen.2012.10.008. Epub 2012 Oct 16. PMID 23079585
- [Background] Rycaj K, Tang DG. Cancer stem cells and radioresistance. Int J Radiat Biol. 2014 Aug;90(8):615-21. doi: 10.3109/09553002.2014.892227. Epub 2014 Mar 7. PMID 24527669

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant Chemoradiation and Surgical Resection: Neoadjuvant chemoradiation: Intensity modulation radiation therapy (IMRT) with a simultaneous integrated boost with Fixed-gantry IMRT, helical tomotherapy, or Vesicular Modulated Arc Therapy (VMAT) can be used. All photon treatments shall be delivered with megavoltage machines of a minimum energy of 6 Megavolt (MV) photons. Selection of the appropriate photon energy(ies) should be based on optimizing the radiation dose distribution within the target volume and minimizing dose to non-target normal tissue.
  Drug Therapy with Temozolomide (benzolamide) (Standard of Care): During Concomitant Radiation Therapy on the same day as the first fraction of radiotherapy. Temozolomide will be administered continuously from day 1 of radiotherapy to the last day of radiation at a daily oral dose of 75 mg/m2 for a maximum of 49 days. The drug will be administered orally daily during radiotherapy, as best tolerated by the patient. During weekends without radiotherapy (Saturday and Sunday), the drug will be taken in the morning. The dose will be determined using actual body surface area (BSA) as calculated in square meters at the beginning of the concomitant treatment. The BSA will be calculated from the height obtained at the pretreatment visit. Capsules of temozolomide are available in 5, 20, 100, 140, 180, and 250 mg.
  Surgery post Radiation and Temozolomide (benzolamide): Surgical resection of GBM will be done after radiation and Temozolomide treatment.
Period: Overall Study
Arm/Group | Neoadjuvant Chemoradiation and Surgical Resection
Started | 2
Completed | 1
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Chemoradiation and Surgical Resection
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: No Study Related Undue Toxicity or Progression
Description: Number of participants with no study related undue toxicity or progression within the limits of stage one patients. Toxicity is defined as: progression precluding surgery, unanticipated neurological decompensation, non-completion of neoadjuvant therapy (other than protocol defined dose adjustments or discontinuation), treatment related delay of >6 weeks to surgery, and/or major unforeseen surgical complication requiring repeat surgical intervention including other than non-life-threatening infection like meningitis/encephalitis or septicemia.
Time Frame: 7 months for each patient from registration
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemoradiation and Surgical Resection
Number analyzed (Participants) | 2
Participants | 2

2. Primary Outcome: Progression Free Survival
Description: Number of participants with Progression Free Survival/clinical progression with new or worsening neurological symptoms related to the tumor and not due to non-tumor or study related symptoms.
Time Frame: 7 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemoradiation and Surgical Resection
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 years
Arm/Group | Neoadjuvant Chemoradiation and Surgical Resection
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemoradiation and Surgical Resection (N=2)
Grade 1 Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Grade 1 Dermatitis (Blood and lymphatic system disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Decrease in blood platelet count (Blood and lymphatic system disorders) | 2 (2)
Grade 3 Lymphocyte decrease (Blood and lymphatic system disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Infection (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT04209790/Prot_SAP_000.pdf